CLINICAL TRIAL: NCT05423652
Title: Aiding COPD and CHF Ultrasound-guided Management Through ENhanced Point Of Care UltraSound
Acronym: ACCUMEN-POCUS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle Grinman (Other)
Collaborators: PRESUNA (Unknown); Institute of Health Economics, Canada (Other); Alberta Boehringer Ingelheim Collaboration (Unknown)
Responsible Party: Sponsor-Investigator, Michelle Grinman, Principal Investigator, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: REB22-0434
Record Dates: First submitted 2022-05-05; First posted 2022-06-21 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: COPD; CHF; Pneumonia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pneumonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POCUS-PRESUNA (Experimental): Daily home hospital care will be enhanced by lung POCUS acquired remotely by community paramedics or in-person by physicians, and interpreted by physicians. They will then document their findings on PRESUNA to obtain a longitudinal record that enables monitoring of trends to support clinical decision-making.
  Interventions: Device: Lung point of care ultrasound; Other: PRESUNA software
- Standard Care (No Intervention): Standard home hospital care

INTERVENTIONS:
Device: Lung point of care ultrasound — Point of care ultrasound of the lungs will be performed to enhance physical assessments as needed to make clinical decisions for patients with CHF, COPD and/or pneumonia. The majority of images will be acquired and uploaded to a web-based portal by community paramedics in patients' homes and interpreted remotely by hospital-based physicians on call for the home hospital.
  Other Names: POCUS
  Arms: POCUS-PRESUNA
Other: PRESUNA software — PRESUNA is a new medical software that enables clinicians to summarize POCUS findings and document them on a platform that provides a visual summary of findings over time. PRESUNA also provides POCUS educators and learners to see the learners' progress over time in terms of the accuracy of their assessments when compared to POCUS experts providing longitudinal mentorship.
  Arms: POCUS-PRESUNA

SUMMARY:
Single-center, two-arm, parallel, randomized controlled trial comparing enhanced daily assessments for patients with COPD and/or CHF using point of care ultrasound with PRESUNA software (POCUS-PRESUNA) versus standard care provided by home-based acute care through a tertiary acute care medical teaching hospital. The objectives are to evaluate POCUS-PRESUNA on improving patient experience, provider experience, improve healthcare utilization/costs, and to test the feasibility of incorporating longitudinal POCUS assessments in home-based acute care via remotely acquired images by non-physicians.

DETAILED DESCRIPTION:
PRESUNA, a new medical software platform that supports clinicians in optimizing their use of POCUS for CHF and COPD patients in the community, is designed to enhance clinical decision-making and long-term monitoring of patients with CHF and COPD. The aim is to more precisely identify changes in the lungs in order to proactively treat exacerbations and confirm treatment responses. It will also enable practitioners to share information from each scan visually and in a standard format in order to track changes longitudinally. This is expected to reduce potentially avoidable hospitalizations and increase patient quality of life in the community.

This study will implement the use of POCUS enhanced by PRESUNA software in the clinical practice of clinicians on a home hospital (HH) program at a tertiary teaching hospital in Calgary, Alberta. On this home hospital, patients are seen and examined either by home visiting community paramedics who consult with the physician, or in-person by physicians in the home hospital clinic space when expedited diagnostic imaging or investigations are required.

Objective:

To perform a randomized control trial comparing patients with COPD and/or CHF admitted to the HH who will undergo usual care versus usual care enhanced with POCUS and PRESUNA.

Methods:

1. Practitioner Recruitment Home hospital clinicians will be provided information about this study in order to obtain informed consent for participation in the study. Physicians who are already POCUS experts will provide informed consent to undergo training on how to use PRESUNA software and to incorporate POCUS into their home hospital care for intervention study patients. Non-POCUS expert clinicians (community paramedics, some of the physicians and nurses) will provide informed consent to undergo group POCUS training and subsequent individual training sessions in order to enable them to become proficient at using POCUS. They will also consent to being trained on how to use PRESUNA software, as well as incorporating POCUS and PRESUNA into their home hospital care for intervention arm patients.
2. Patient Recruitment Patients admitted to HH with CHF and/or COPD will be approached to participate in the research study by the Nurse Navigator or Research Assistant. Those that provide informed consent will be randomized (1:1) to the intervention (POCUS-PRESUNA enhanced HH care) versus control group (usual HH care).

ELIGIBILITY:
Patient Inclusion Criteria:

* 18 years of age or older
* Has a provincial health care number
* Functionally safe to receive HH care or have sufficient caregiving to support them at home
* Stable enough to be cared for at home - stable vital signs and requiring no more than 2 visits per day
* Able and willing to follow a management plan
* Provides consent to receive care on HH
* Diagnosis of CHF and/or COPD that requires HH care
* No painful/broken ribs that could be affected by pressure applied when performing lung POCUS

Patient Exclusion Criteria:

* Not eligible for HH care
* New unstable rib fractures
* Prior history of allergy to ultrasound gel
* Participant refusal to participate in research study

Provider inclusion criteria

* Attending clinician on the home hospital program within the next 3-6 months
* Provides informed consent to participate in the study, including necessary training for the use of POCUS and/or PRESUNA

Provider exclusion criteria

* Not a home hospital clinician
* Refuses to consent for the study / training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Length of stay | From the date of admission to discharge from the index admission, assessed up to 1 year
  Length of stay for index Home Hospital admission

SECONDARY OUTCOMES:
Patient outcome - Time to resolution of infection | Assessed up to 24 months after infection identified
  return to baseline oxygen saturation and normalization of white blood cell count
Patient outcome - time to decongestion | Assessed up to one year after congestion identified
  absence of crackles and baseline oxygen saturation on lung examination
Patient outcome - rate of change in NT-BNP | Change from admission to when decongestion occurred, assessed up to 12 months
  Difference between NT-BNP on admission and at time of decongestion over total number of days
Patient outcome - Admission to facility living | From date and time of discharge from index admission, assessed up to 12 months
  Proportion of patients in each study arm that required admission to facility living (eg: long-term care, supportive living) after their index admission
Patient outcome - Escalation of care | From date of randomization until the patient is discharged from the index admission (assessed up to 12 months).
  Incidence rate ratio for frequency with which patients are transferred back to the bricks and mortar hospital from the home hospital.
Patient outcome - Adverse events | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first until the patient is discharged from the hospital (assessed up to 12 months).
  Frequency and severity of adverse events (venous thromboembolism, new infections, falls, delirium)
Patient outcome - Mortality | From date of randomization until the date of death, assessed up to 12 months
  Date and cause of mortality of occurrence of mortality
Health Related Quality of Life - EuroQuol- 5-Dimension-5-Level (EQ-5D-5L) -Mobility | At time of randomization, within one week of discharge from the index admission, at 3 months post-discharge, and at 6 months post-discharge
  The ability to mobilize is rated by patients on a scale from 1-5 (1= no problems, 2= slight problems, 3= moderate problems, 4= Severe problems, 5= Unable to perform activity)
Health Related Quality of Life - EuroQuol- 5-Dimension-5-Level (EQ-5D-5L) -Activities of daily living | At time of randomization, within one week of discharge from the index admission, at 3 months post-discharge, and at 6 months post-discharge
  Ability to perform activities of daily living rated by patients from 1-5 (1= no problems, 2= slight problems, 3= moderate problems, 4= Severe problems, 5= Unable to perform activity)
Health Related Quality of Life - EuroQuol- 5-Dimension-5-Level (EQ-5D-5L) -Pain and discomfort | At time of randomization, within one week of discharge from the index admission, at 3 months post-discharge, and at 6 months post-discharge
  The intensity of pain or discomfort is rated by patients from 1 to 5 (1=none, 2= slight , 3= moderate , 4=severe, 5=extreme).
Health Related Quality of Life - EuroQuol- 5-Dimension-5-Level (EQ-5D-5L) -Self care | At time of randomization, within one week of discharge from the index admission, at 3 months post-discharge, and at 6 months post-discharge
  Ability to perform self-care rated from 1= no problems, 2= slight problems, 3= moderate problems, 4= Severe problems, 5= Unable to perform activity
Health Related Quality of Life - EuroQuol- 5-Dimension-5-Level (EQ-5D-5L) -Anxiety and Depression | At time of randomization, within one week of discharge from the index admission, at 3 months post-discharge, and at 6 months post-discharge
  Patients rate whether they feel anxious or depressed from 1-5 (1=no, 2= slightly, 3= moderately, 4=severely, 5=extremely).
Health Related Quality of Life - EuroQuol- 5-Dimension-5-Level (EQ-5D-5L) -Index Score | At time of randomization, within one week of discharge from the index admission, at 3 months post-discharge, and at 6 months post-discharge
  The index score is computed using the EQ-5D calculator that uses the scores of the individual dimensions (mobility, self-care, activities of daily living, pain and discomfort, anxiety and depression); Scores range between 5-25 with higher scores indicating a worse outcome
Health Related Quality of Life - EuroQuol- 5-Dimension-5-Level (EQ-5D-5L) Visual Analogue Scale (EQ-VAS) | At time of randomization, within one week of discharge from the index admission, at 3 months post-discharge, and at 6 months post-discharge
  Participant asked to rate both verbally and visually "where [they] would put [their] health today" on a scale from 0 ("the worst health you can imagine") to 100 ("the best health you can imagine)
Patient experience | Upon discharge from the Home Hospital (up to 7 business days post-discharge)
  Survey measuring experience with clinical care and various technologies employed by the Home Hospital (digital remote patient monitoring, videoconferencing, as well as POCUS for the intervention arm). This survey was developed by the study team. Responses to questions were either, "yes", "yes, to some extent", "no", and "unsure".
Provider experience | Within 1 week of being on the Hospital at Home service
  Surveys including experience providing care for patients on each study arm and experience with various technologies employed in the home hospital program (digital remote patient monitoring, videoconferencing, as well as POCUS and PRESUNA for the intervention arm). This survey was developed by the study team. Responses were on a Likert scale, which included "strongly disagree", "disagree", "neither agree/nor disagree", "agree" and "strongly agree"
Healthcare utilization cost - Diagnostic testing | Between the date and time of hospital admission to up to 3 months post-discharge
  Cost of Diagnostic testing
Healthcare utilization - Incidence rate ratio of acute care days pre/during/post | 90 days before randomization until 90 days after index admission (assessed up to 15 months)
  Incidence rate ratio of acute care days in the bricks and mortar hospital 90 days pre-randomization, during the index admission after randomization, and 90 days post discharge from index admission
Healthcare utilization - Incidence rate ratio of ED/Urgent Care visits pre/during/post | 90 days before, during and 90 days after index admission
  Incidence rate ratio of ED and urgent care visits- 90 days pre-randomization, during the index admission after randomization, and 90 days post discharge from index admission
Cost analysis | From date of admission until the date of discharge from the index admission, assessed up to 12 months").
  Incremental effectiveness ratio for the index admission
Cost analysis | From date of discharge from index admission, assessed up to 90 days.
  Incremental effectiveness ratio for healthcare utilization post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Grinman, MD FRCPC MPH, Principal Investigator — University of Calgary
Locations (1):
- Rockyview General Hospital, Calgary, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grinman MN, Nakhla P, Reid S, Moon D, Dehghan Noudeh N, Olaosebikan O, Ip ACY, Saunders S, Kozicky R, Conly J, Kirkpatrick AW, Round J, Ma IWY, Pascoe S, Altabbaa G. Aiding Chronic Obstructive Pulmonary Disease and Congestive Heart Failure Ultrasound-Guided Management Through Enhanced Point-of-Care Ultrasound (ACCUMEN-POCUS): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 23;14:e76186. doi: 10.2196/76186. PMID 40987446